CLINICAL TRIAL: NCT03190343
Title: Assessment of Cholangio-pancreatoscopy for the Diagnosis and the Treatment of Biliary and Pancreatic Diseases Trial " EASYSPY "
Brief Title: Assessment of Cholangio-pancreatoscopy for the Diagnosis and the Treatment of Biliary and Pancreatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, Arthur Laquiere, Gastroenterologist, Hospital St. Joseph, Marseille, France
Other Study IDs: CCTIRS 16-351
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Lesions of Biliary or Wirsung Ducts; Biliary Tract Diseases; Common Bile Duct Diseases; Pancreatic Duct Disorder
MeSH Terms: conditions — Biliary Tract Diseases; Common Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cholangio-pancreatoscopy

SUMMARY:
The biliary and pancreatic tumors are rare but the prognosis is pejorative. It was difficult to have histology of these tumors as the samples taken during ERCP were performed under " blind " radiology control. So the diagnostic accuracy was insufficient.

The arrival of A new optic fiber endoscope used by only one operator had improved the diagnostic of bilio-pancreatic diseases. However this technology with optic fiber quickly had proved outdated for several reasons: poor manoeuvrability, perfectible optical vision, optical fibers fragility and cost.

A new generation of endoscopes with digital vision appeared and would allow an increase in diagnostic accuracy related to better vision and manoeuvrability.

The purpose of the study is to assess the interest of the cholangio pancreatoscopy performed with digital vision.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with biliary duct stenosis with undetermined etiology
* Patients with pancreatic duct stenosis with undetermined etiology
* Patients with pancreatic duct distension with undetermined etiology
* Patients with biliary or pancreatic gallstones after failure to endoscopic treatment

Exclusion Criteria:

* Patients with haemorrhagic disease or hemostasis and coagulation disorders (TP < 60%, TCA> 40 sec. and platelets < 60000/mm3).
* Patients treated with anticoagulant or platelet aggregation inhibiting drugs that could not be temporarily interrupted.
* Patients with biliary duct diameter < 3 mm
* Patients with pancreatic duct diameter <3 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENTS WITH BILIARY OR PANCREATIC DUCT STENOSIS
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic accuracy of the Spyglass to distinguish a benign lesion from a malignant lesion of the biliary or Wirsung ducts. | 4 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: ARTHUR LAQUIERE, MD, Principal Investigator — French Society of Digestive Endoscopy
Locations (3):
- France (3):
  - Hopital Mermoz, Lyon
  - Hopital Saint Joseph, Marseille
  - Centre Hospitalier Jacques Lacarin, Vichy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nakeeb A, Pitt HA, Sohn TA, Coleman J, Abrams RA, Piantadosi S, Hruban RH, Lillemoe KD, Yeo CJ, Cameron JL. Cholangiocarcinoma. A spectrum of intrahepatic, perihilar, and distal tumors. Ann Surg. 1996 Oct;224(4):463-73; discussion 473-5. doi: 10.1097/00000658-199610000-00005. PMID 8857851
- [Result] Bar-Meir S, Rotmensch S. A comparison between peroral choledochoscopy and endoscopic retrograde cholangiopancreatography. Gastrointest Endosc. 1987 Feb;33(1):13-4. doi: 10.1016/s0016-5107(87)71476-x. PMID 3557026
- [Result] Tringali A, Lemmers A, Meves V, Terheggen G, Pohl J, Manfredi G, Hafner M, Costamagna G, Deviere J, Neuhaus H, Caillol F, Giovannini M, Hassan C, Dumonceau JM. Intraductal biliopancreatic imaging: European Society of Gastrointestinal Endoscopy (ESGE) technology review. Endoscopy. 2015 Aug;47(8):739-53. doi: 10.1055/s-0034-1392584. Epub 2015 Jul 6. PMID 26147492
- [Result] Urakami Y, Seifert E, Butke H. Peroral direct cholangioscopy (PDCS) using routine straight-view endoscope: first report. Endoscopy. 1977 Mar;9(1):27-30. doi: 10.1055/s-0028-1098481. PMID 862583
- [Result] Ramchandani M, Reddy DN, Gupta R, Lakhtakia S, Tandan M, Darisetty S, Sekaran A, Rao GV. Role of single-operator peroral cholangioscopy in the diagnosis of indeterminate biliary lesions: a single-center, prospective study. Gastrointest Endosc. 2011 Sep;74(3):511-9. doi: 10.1016/j.gie.2011.04.034. Epub 2011 Jul 7. PMID 21737076
- [Result] Draganov PV, Lin T, Chauhan S, Wagh MS, Hou W, Forsmark CE. Prospective evaluation of the clinical utility of ERCP-guided cholangiopancreatoscopy with a new direct visualization system. Gastrointest Endosc. 2011 May;73(5):971-9. doi: 10.1016/j.gie.2011.01.003. Epub 2011 Mar 17. PMID 21419408
- [Result] Rey JW, Hansen T, Dumcke S, Tresch A, Kramer K, Galle PR, Goetz M, Schuchmann M, Kiesslich R, Hoffman A. Efficacy of SpyGlass(TM)-directed biopsy compared to brush cytology in obtaining adequate tissue for diagnosis in patients with biliary strictures. World J Gastrointest Endosc. 2014 Apr 16;6(4):137-43. doi: 10.4253/wjge.v6.i4.137. PMID 24748921
- [Result] Navaneethan U, Hasan MK, Lourdusamy V, Njei B, Varadarajulu S, Hawes RH. Single-operator cholangioscopy and targeted biopsies in the diagnosis of indeterminate biliary strictures: a systematic review. Gastrointest Endosc. 2015 Oct;82(4):608-14.e2. doi: 10.1016/j.gie.2015.04.030. Epub 2015 Jun 10. PMID 26071061
- [Result] Boyer J. [Endoscopic sphincterotomy and lithiasis of the common bile duct. Reality and perspectives]. Gastroenterol Clin Biol. 1993;17(4):241-3. No abstract available. French. PMID 8339881
- [Result] Seelhoff A, Schumacher B, Neuhaus H. Single operator peroral cholangioscopic guided therapy of bile duct stones. J Hepatobiliary Pancreat Sci. 2011 May;18(3):346-9. doi: 10.1007/s00534-010-0360-7. PMID 21480000
- [Result] Arnelo U, Siiki A, Swahn F, Segersvard R, Enochsson L, del Chiaro M, Lundell L, Verbeke CS, Lohr JM. Single-operator pancreatoscopy is helpful in the evaluation of suspected intraductal papillary mucinous neoplasms (IPMN). Pancreatology. 2014 Nov-Dec;14(6):510-4. doi: 10.1016/j.pan.2014.08.007. Epub 2014 Sep 27. PMID 25287157
- [Derived] Laquiere AE, Privat J, Fumex F, Grandval P, Lecomte L, Curel L, Belle A, Trottier-Tellier F, Urena-Campos R, Penaranda G, Boustiere C, Napoleon B. Performance of digital single-operator cholangiopancreatoscope for biliopancreatic diseases in real life: results from a prospective multicenter study. Scand J Gastroenterol. 2020 Nov;55(11):1381-1388. doi: 10.1080/00365521.2020.1832143. Epub 2020 Oct 23. PMID 33095075